CLINICAL TRIAL: NCT04361019
Title: Physical Activity in University Students Around COVID-19 Confinement: Determinants and Consequences on Health Status and Quality of Life
Brief Title: Physical Activity in University Students Around COVID-19 Confinement
Status: Completed | Type: Observational
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Collaborators: University of Cadiz (Other); University of Extremadura (Other); Universidad de Zaragoza (Other); Universidad de Granada (Other); University of Castilla-La Mancha (Other); University of Las Palmas de Gran Canaria (Other); Universidad de León (Other); University of Seville (Other); University of Valencia (Other); Universidad Miguel Hernandez de Elche (Other); Technical University of Madrid (Other); Universidad Pública de Navarra (Other); University of the Balearic Islands (Other); Universitat Jaume I (Other); University of Cantabria (Other)
Responsible Party: Principal Investigator, Jon Irazusta, Dr, University of the Basque Country (UPV/EHU)
Other Study IDs: Covid_PA2020
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Physical Activity
Keywords: University Students; Survey; COVID-19; Confinement; Physical Activity; Quality of Life; Health; Sleep; Pain
MeSH Terms: conditions — Motor Activity; COVID-19; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: On-Line Survey — A survey has been sent by email to the students of the participating universities

SUMMARY:
The period of confinement due to COVID-19 may lead to reduced physical activity levels with negative consequences for health and quality of life in the short and long term, in case the sedentary habits are maintained over time. It is therefore essential to know the physical activity and health habits of university students during the confinement, as it could help in the design of effective strategies for the post-confinement period, as well as for any similar future situations. The general objective of the study is to know how university students have adapted their physical activity and health habits to the situation of confinement generated by COVID-19, as well as to identify the determining factors and the possible consequences. It is expected that there will be modifications in the patterns of physical activity in this situation, which could vary based on sociodemographic and economic determinants, and could affect parameters of health and quality of life. A survey will be sent to all students by email through the corresponding vice-rectorates of the sixteen participating universities (https://covid19.ehu.es/). The survey will be completed "online" anonymously. Among those participants who wish to keep participating in the study, a follow-up will be carried out one month and one year after the end of the confinement period. In this case, those subjects must indicate their willingness to keep participating and provide a contact email. The follow-up period will allow to know how physical activity and health habits are modified in the long term.

ELIGIBILITY:
Inclusion Criteria:

* University students of any degree (bachellor's degree, master's degree, doctorate degree or any other University studies

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All University students from the 16 Universities participating in the study will be invited to answer the online survey. The total amount of students in the 16 universities is around 500,000. The sample will include students in different academic degrees: bachelor's degree, master's degree, doctorate degree or any other University studies.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
: International Physical Activity Questionnaire - Short Form | April-May, 2020
  7-item questionnaire regarding last 7 days' physical activity and sedentary behavior. Vigorous, moderate and walking physical activities will be measured in METS (metabolic equivalent of task) per week, and sedentary behavior will be collected as sedentary time per day
: International Physical Activity Questionnaire - Short Form | June 2020
  7-item questionnaire regarding last 7 days' physical activity and sedentary behavior. Vigorous, moderate and walking physical activities will be measured in METS (metabolic equivalent of task) per week, and sedentary behavior will be collected as sedentary time per day
: International Physical Activity Questionnaire - Short Form | April-May, 2021
  7-item questionnaire regarding last 7 days' physical activity and sedentary behavior. Vigorous, moderate and walking physical activities will be measured in METS (metabolic equivalent of task) per week, and sedentary behavior will be collected as sedentary time per day

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index: Subjective Sleep Quality and Sleep Duration domains | April-May, 2020
  19-item self-report questionnaire assessing 7 domains regarding sleep. Only item number 4 (corresponding to subjective sleep quality domain) and item number 6 (corresponding to sleep duration domain) will be measured
Pittsburgh Sleep Quality Index: Subjective Sleep Quality and Sleep Duration domains | June, 2020
  19-item self-report questionnaire assessing 7 domains regarding sleep. Only item number 4 (corresponding to subjective sleep quality domain) and item number 6 (corresponding to sleep duration domain) will be measured
Pittsburgh Sleep Quality Index: Subjective Sleep Quality and Sleep Duration domains | April-May, 2021
  19-item self-report questionnaire assessing 7 domains regarding sleep. Only item number 4 (corresponding to subjective sleep quality domain) and item number 6 (corresponding to sleep duration domain) will be measured
Short Form 36 Health Survey: Bodily Pain domain | April-May 2020
  The Short Form 36 Health Survey is a 36 -item self-report questionnaire assessing 8 domains regarding health-related quality of life. Only items number 7 and 8 (corresponding to bodily pain domain) will be measured. A score ranging from 0 to 100 is obtained, with higher scores indicating a better bodily pain related quality of life
Short Form 36 Health Survey: Bodily Pain domain | June, 2020
  The Short Form 36 Health Survey is a 36 -item self-report questionnaire assessing 8 domains regarding health-related quality of life. Only items number 7 and 8 (corresponding to bodily pain domain) will be measured. A score ranging from 0 to 100 is obtained, with higher scores indicating a better bodily pain related quality of life
Short Form 36 Health Survey: Bodily Pain domain | April-May, 2021
  The Short Form 36 Health Survey is a 36 -item self-report questionnaire assessing 8 domains regarding health-related quality of life. Only items number 7 and 8 (corresponding to bodily pain domain) will be measured. A score ranging from 0 to 100 is obtained, with higher scores indicating a better bodily pain related quality of life
EuroQol 5D: Self rated health | April-May, 2020
  The EuroQol 5D is a self-report questionnaire to assess five health-related domains. Only the item assessing the overall self-rated health status will be used. In the traditional questionnaire, participants are asked to rate their current health status in a 0-100 visual analogue scale, with "0" corresponding to "the worst health you can imagine" and "100" to "the best health you can imagine". A modified version using a 0-10 numerical rating scale will be used, in order to adapt it to an online format
EuroQol 5D: Self rated health | June, 2020
  The EuroQol 5D is a self-report questionnaire to assess five health-related domains. Only the item assessing the overall self-rated health status will be used. In the traditional questionnaire, participants are asked to rate their current health status in a 0-100 visual analogue scale, with "0" corresponding to "the worst health you can imagine" and "100" to "the best health you can imagine". A modified version using a 0-10 numerical rating scale will be used, in order to adapt it to an online format
EuroQol 5D: Self rated health | April-May, 2021
  The EuroQol 5D is a self-report questionnaire to assess five health-related domains. Only the item assessing the overall self-rated health status will be used. In the traditional questionnaire, participants are asked to rate their current health status in a 0-100 visual analogue scale, with "0" corresponding to "the worst health you can imagine" and "100" to "the best health you can imagine". A modified version using a 0-10 numerical rating scale will be used, in order to adapt it to an online format

OTHER OUTCOMES:
Sociodemographic outcomes | April-May, 2020
  Sociodemographic variables will include age, gender, height, weight, residence (place and family unit type and size), academic data (University, branch of knowledge and academic degree) and smoking habits
Sociodemographic outcomes | June, 2020
  Sociodemographic variables will include age, gender, height, weight, residence (place and family unit type and size), academic data (University, branch of knowledge and academic degree) and smoking habits
Sociodemographic outcomes | April-May, 2021
  Sociodemographic variables will include age, gender, height, weight, residence (place and family unit type and size), academic data (University, branch of knowledge and academic degree) and smoking habits
COVID-19 related factors | April-May, 2020
  Participants will be asked if: a) they have had COVID-19 related symptoms, b) have been diagnosed with COVID-19 by a health professional or c) have been living with a person diagnosed with COVID-19 during the confinement
COVID-19 related factors | June, 2020
  Participants will be asked if: a) they have had COVID-19 related symptoms, b) have been diagnosed with COVID-19 by a health professional or c) have been living with a person diagnosed with COVID-19 during the confinement
COVID-19 related factors | April-May, 2021
  Participants will be asked if: a) they have had COVID-19 related symptoms, b) have been diagnosed with COVID-19 by a health professional or c) have been living with a person diagnosed with COVID-19 during the confinement

CONTACTS AND LOCATIONS:
Overall Officials: Jon Irazusta, PhD, Principal Investigator — Basque Country University (UPV-EHU), Leioa, Bizkaia, 48940, Spain
Locations (1):
- Basque Country University (UPV-EHU),, Bilbao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Yes
All individual data of the participants, with the exception of the email, the university and where they live, will be available upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available once the study will finish
Access Criteria: The access to individual participant data will be decided after analysing each request taking into account the scientific quality of the proposal

REFERENCES:
- [Background] Bassett DR Jr. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1396. doi: 10.1249/01.MSS.0000078923.96621.1D. No abstract available. PMID 12900695
- [Background] Rodriguez-Munoz S, Corella C, Abarca-Sos A, Zaragoza J. Validation of three short physical activity questionnaires with accelerometers among university students in Spain. J Sports Med Phys Fitness. 2017 Dec;57(12):1660-1668. doi: 10.23736/S0022-4707.17.06665-8. Epub 2017 Mar 1. PMID 28249383
- See also: Link to the online survey used in the study — http://covid19.ehu.es/